CLINICAL TRIAL: NCT04778319
Title: Hysterosalpingography and Hysteroscopy in Intracytoplasmic Sperm Injection
Brief Title: Hysterosalpingography and Hysteroscopy in ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: tubal disease
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tubal occlusion (Active Comparator): occlusion of tubes
  Interventions: Other: occlusion of tubes
- non occlusion of tube (Sham Comparator): non occlusion of tubes
  Interventions: Other: non occlusion of tubes

INTERVENTIONS:
Other: occlusion of tubes — to occlude the fallopian tubes
  Arms: tubal occlusion
Other: non occlusion of tubes — not to occlude the tubes
  Arms: non occlusion of tube

SUMMARY:
unexplained infertility is a rising problem in clinical practice

DETAILED DESCRIPTION:
Assessment of uterine cavity is very important before ICSI

ELIGIBILITY:
Inclusion Criteria:

* women with infertility

Exclusion Criteria:

* women with medical disorders

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with infertility
Enrollment: 200 (Estimated)
Dates: Start 2021-03-02 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
the number of women who will become pregnant | 3 months
  number of women who will have positive pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt